CLINICAL TRIAL: NCT03049436
Title: Adapted Physical Activity in a Chemotherapy Ambulatory Care Unit: Feasibility and Impact on Fatigue, Anxiety and Depression in Cancer Patients
Acronym: UMACHAPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ17008
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-01

CONDITIONS: Adapted Physical Activity and Cancer
Keywords: Physical activity; cancer; chemotherapy; daily care unit
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with program of adapted physical activity
  Interventions: Other: Program of adapted physical activity

INTERVENTIONS:
Other: Program of adapted physical activity

SUMMARY:
Physical activity has demonstrated efficacy in cancer prevention and improves quality of life and outcome in cancer survivors. Patients undergoing chemotherapy, especially those with advanced disease, may have symptoms leading to inactivity. Adapted physical activity (APA) among those patients could improve their tolerance to the treatment, and thereby their quality of life. APA could be beneficial to patients with curable disease as well as patients undergoing palliative chemotherapy. Some studies suggest that fighting against loss of muscle mass could lead to a survival benefit. However, APA is not established in daily practice and has not yet been evaluated in a chemotherapy ambulatory care unit.

Primary aim of the study is to assess feasibility of an APA program in a chemotherapy ambulatory care unit of digestive, lung, hematological and dermatological cancers Secondary aim is to measure the impact of an APA program on fatigue, anxiety, depression and handgrip strength in patients beginning chemotherapy or targeted therapy for a digestive, lung, hematological or dermatological cancer, of any stage.

DETAILED DESCRIPTION:
Assess feasibility of an APA program in a chemotherapy ambulatory care unit of digestive, lung, hematological, and dermatological cancers Measure the impact of an APA program on fatigue, anxiety, depression, handgrip strength

ELIGIBILITY:
Inclusion Criteria:

* Patients beginning chemotherapy or targeted therapy at UMA-CH ambulatory care unit of Reims, CHU, for a digestive, lung, hematological or dermatological cancer, of any stage
* Patients who agree to participate to the study
* Major patient

Exclusion Criteria:

* Patient with previous chemotherapy or targeted therapy in the UMA-CH unit
* Patient under law protection
* Minor patient
* Patient with neurological defect preventing from any physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing chemotherapy or targeted therapy at UMA-CH ambulatory care service of Reims, CHU, for a digestive, lung, hematological or dermatological cancers, of any stage, between February 2017 and August 2017
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of APA program | Day 0
  Percentage of patients accepting APA program

SECONDARY OUTCOMES:
fatigue | Month 3
  Fatigue evaluating using the Multidimensional Fatigue Inventory. The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument assessing the following items: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. It has been validated to assess fatigue in cancer patients.
Anxiety | Month 3
  Anxiety evaluating using Hospital Anxiety and Depression scale. Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression, in a two factors model, without confounding with somatic or psychiatric disorders, and has been validated in cancer patients.
Fatigue | Month 6
  Fatigue evaluating using the Multidimensional Fatigue Inventory. The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument assessing the following items: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.
Anxiety | Month 6
  Anxiety evaluating using Hospital Anxiety and Depression scale. Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression, in a two factors model, without confounding with somatic or psychiatric disorders, and has been validated in cancer patients.
handgrip strength | Month 3
  handgrip strength evaluating using Hand grip test. Hand grip test allows the measurement of muscle strength of the upper limbs, which is a reflection of the overall strength of an individual. Thresholds for the loss of muscle strength are <17kg in women and <30 kg in men.
handgrip strength | Month 6
  handgrip strength evaluating using Hand grip test. Hand grip test allows the measurement of muscle strength of the upper limbs, which is a reflection of the overall strength of an individual. Thresholds for the loss of muscle strength are <17kg in women and <30 kg in men.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France